CLINICAL TRIAL: NCT05831475
Title: Leveraging Exercise to Age in Place (LEAP) Together: An Intergenerational Intervention to Address Loneliness and Social Isolation
Brief Title: LEAPTogether: An Intergenerational Intervention to Address Loneliness and Social Isolation
Acronym: LEAPTogether
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: FlexTogether (Unknown)
Responsible Party: Principal Investigator, Allison Mays, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001980
Record Dates: First submitted 2023-02-06; First posted 2023-04-26 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Social Isolation; Loneliness; Intergenerational Relations
Keywords: physical activity; older adults; intergenerational; social isolation; loneliness; virtual exercise
MeSH Terms: conditions — Social Isolation; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be randomized by the coordinator to a study arm:
  Arm 1- older adult paired with older adult (40) Arm 2- older adult paired with younger adult (20 older, 20 younger)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer Pairings (Experimental): Two older adults paired
  Interventions: Behavioral: Peer Virtual Paired Exercise
- Intergenerational Pairings (Experimental): A younger adult and older adult paired
  Interventions: Behavioral: Intergenerational Virtual Paired Exercise

INTERVENTIONS:
Behavioral: Intergenerational Virtual Paired Exercise — Participants will be paired with someone older/ younger and will engage in exercise videos with the ability to simultaneously video chat with their partner while exercising. Participants will log on with their partner twice a week for 8 weeks.
  Arms: Intergenerational Pairings
Behavioral: Peer Virtual Paired Exercise — Participants will be paired with someone of the same age group and will engage in exercise videos with the ability to simultaneously video chat with their partner while exercising. Participants will log on with their partner twice a week for 8 weeks.
  Arms: Peer Pairings

SUMMARY:
Older adult participants will engage in exercise videos twice a week for 8 weeks either while paired with a peer (same age group) or paired with a younger adult with the ability to simultaneously video chat while exercising.

DETAILED DESCRIPTION:
Participation in this study includes:

* Completing assessments at baseline (start of study), 8 weeks, and 16 weeks
* Initial meeting with an Exercise Physiologist to determine exercise interests and preferences
* Being matched with an exercise partner
* Virtually meeting with partner to engage in exercise videos via the FlexTogether platform (meet twice a week for a total of 8 weeks)
* Attend a live group class once a month
* Completing an exit interview

Primary Objective:

To assess feasibility by monitoring adherence to an 8-week virtual paired exercise program for older adults

Secondary Objectives:

1. To mechanistically investigate the key social pairing components (i.e., older adults together, younger and older adult pairing) within a virtual program necessary to enhance social connectedness, decrease loneliness, improve well-being, and increase physical activity in older adults and younger adult participants in the short-term (pre-post) through surveys and qualitative interviews
2. To mechanistically investigate the key social pairing components (i.e., older adults together, younger and older adult pairing) within a virtual program necessary to enhance social connectedness, decrease loneliness, improve well-being, and increase physical activity in older adults and younger adult participants in the long-term (8 weeks post-intervention / 18 weeks on study) through surveys and qualitative interviews

ELIGIBILITY:
Inclusion Criteria:

* Verbal informed consent obtained from subject and ability for subject to comply with the requirements of the study
* Age 18-30 years for younger adults
* Age greater than or equal to 65 years for older adults
* Has access to a tablet, laptop, or desktop computer with video capabilities connected to the internet with a screen at least 13 inches across
* Able to read, write, and understand English
* Has a 5 x 6 foot space at home in which to exercise

Exclusion Criteria:

* Current diagnosis of dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Adherence to an 8-week virtual paired exercise program for older adults | Attendance over 8-weeks
  Adherence defined as attending at least 12 out of 16 sessions (70% attendance)

SECONDARY OUTCOMES:
social connectedness per units in scale | baseline and 10 weeks
  To mechanistically investigate the key social pairing components (i.e. solo, older adults together, younger and older adult pairing) within a virtual program necessary to enhance social connectedness in the short-term (pre-post) through Duke Social Support Index (min score- 11, max score- 33; higher score indicates higher social support and interaction).
pre/post loneliness per units in scale | baseline and 10 weeks
  To mechanistically investigate the key social pairing components (i.e. solo, older adults together, younger and older adult pairing) within a virtual program necessary to decrease loneliness in the short-term (pre-post) through UCLA Loneliness Survey (min score- 3, max score- 9; higher scores correspond to higher feelings of loneliness)
pre/post emotional, social, and psychological well-being per units in scale | baseline and 10 weeks
  To mechanistically investigate the key social pairing components (i.e. solo, older adults together, younger and older adult pairing) within a virtual program necessary to improve well-being in the short-term (pre-post) through Mental Health Continuum Short-Form (min score- 14, max score- 84; higher scores indicate greater levels of positive well-being)
pre/post expectations regarding aging per units in scale | baseline and 10 weeks
  To mechanistically investigate the key social pairing components (i.e. solo, older adults together, younger and older adult pairing) within a virtual program necessary to improve well-being in the short-term (pre-post) through Expectations Regarding Aging Survey (min score- 12, max score- 48; higher score indicates higher (positive) expectations of aging)
pre/post generativity per units in scale | baseline and 10 weeks
  To mechanistically investigate the key social pairing components (i.e. solo, older adults together, younger and older adult pairing) within a virtual program necessary to improve well-being in the short-term (pre-post) through Baltimore Experience Corps Trial Generativity Scale (min score- 13, max score- 65; higher score indicates higher levels of generativity)
pre/post physical activity per units in scale | baseline and 10 weeks
  To mechanistically investigate the key social pairing components (i.e. solo, older adults together, younger and older adult pairing) within a virtual program necessary to increase physical activity in older adults and younger adult participants in the short-term (pre-post) through Godin Leisure Time Exercise Questionnaire (min score- 0, max score- 24+; total of 14 or less indicates insufficient activity/sedentary lifestyle, 24 units or more indicates active lifestyle)
pre/post physical activity per 30 second sit to stand | baseline and 10 weeks
  To mechanistically investigate the key social pairing components (i.e. solo, older adults together, younger and older adult pairing) within a virtual program necessary to increase physical activity in older adults and younger adult participants in the short-term (pre-post) through 30 second sit to stand (how many times can the participant sit and stand without using their hands in a 30 second period, higher number indicates higher level of endurance)
long-term social connectedness per units in scale | 18 weeks
  To mechanistically investigate the key social pairing components (i.e. solo, older adults together, younger and older adult pairing) within a virtual program necessary to enhance social connectedness in the long-term (4.5 months/18 weeks) through Duke Social Support Index (min score- 11, max score- 33; higher score indicates higher social support and interaction).
long-term loneliness per units in scale | 18 weeks
  To mechanistically investigate the key social pairing components (i.e. solo, older adults together, younger and older adult pairing) within a virtual program necessary to decrease loneliness in the long-term (4.5 months/18 weeks) through UCLA Loneliness Survey (min score- 3, max score- 9; higher scores correspond to higher feelings of loneliness)
long-term expectations regarding aging per units in scale | 18 weeks
  To mechanistically investigate the key social pairing components (i.e. solo, older adults together, younger and older adult pairing) within a virtual program necessary to improve well-being in the long-term (4.5 months/18 weeks) through Expectations Regarding Aging Survey (min score- 12, max score- 48; higher score indicates higher (positive) expectations of aging)
long-term emotional, social, and psychological well-being per units in scale | 18 weeks
  To mechanistically investigate the key social pairing components (i.e. solo, older adults together, younger and older adult pairing) within a virtual program necessary to improve well-being in the long-term (4.5 months/18 weeks) through Mental Health Continuum Short-Form (min score- 14, max score- 84; higher scores indicate greater levels of positive well-being)
long-term generativity per units in scale | 18 weeks
  To mechanistically investigate the key social pairing components (i.e. solo, older adults together, younger and older adult pairing) within a virtual program necessary to improve well-being in the long-term (4.5 months/18 weeks) through Baltimore Experience Corps Trial Generativity Scale (min score- 13, max score- 65; higher score indicates higher levels of generativity)
long-term physical activity per units in scale | 18 weeks
  To mechanistically investigate the key social pairing components within a virtual program necessary to increase physical activity in older adults and younger adult participants in the long-term (4.5 months/18 weeks) through Godin Leisure Time Exercise Questionnaire (min score- 0, max score- 24+; total of 14 or less indicates insufficient activity/sedentary lifestyle, 24 units or more indicates active lifestyle)
long-term physical activity per 30 second sit to stand | 18 weeks
  To mechanistically investigate the key social pairing components within a virtual program necessary to increase physical activity in older adults and younger adult participants in the long-term (4.5 months/18 weeks) through 30 second sit to stand (how many times can the participant sit and stand without using their hands in a 30 second period, higher number indicates higher level of endurance)
Key social pairing components in virtual programming | 10 weeks
  Qualitative interview to capture any other thoughts and observations from participants that are not easily captured in surveys

CONTACTS AND LOCATIONS:
Overall Officials: Celina H Shirazipour, Ph.D., Principal Investigator — Cedars-Sinai Medical Center; Allison M Mays, MD, MAS, Principal Investigator — Cedars-Sinai Medical Center; Sonja Rosen, MD, FACP, AGSF, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Beverly Hills, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steptoe A, Shankar A, Demakakos P, Wardle J. Social isolation, loneliness, and all-cause mortality in older men and women. Proc Natl Acad Sci U S A. 2013 Apr 9;110(15):5797-801. doi: 10.1073/pnas.1219686110. Epub 2013 Mar 25. PMID 23530191
- [Background] Tiwari SC. Loneliness: A disease? Indian J Psychiatry. 2013 Oct;55(4):320-2. doi: 10.4103/0019-5545.120536. No abstract available. PMID 24459300
- [Background] Perissinotto CM, Stijacic Cenzer I, Covinsky KE. Loneliness in older persons: a predictor of functional decline and death. Arch Intern Med. 2012 Jul 23;172(14):1078-83. doi: 10.1001/archinternmed.2012.1993. PMID 22710744
- [Background] Ronzi S, Orton L, Pope D, Valtorta NK, Bruce NG. What is the impact on health and wellbeing of interventions that foster respect and social inclusion in community-residing older adults? A systematic review of quantitative and qualitative studies. Syst Rev. 2018 Jan 30;7(1):26. doi: 10.1186/s13643-018-0680-2. PMID 29382375
- [Background] Teater B. Intergenerational Programs to Promote Active Aging: The Experiences and Perspectives of Older Adults. Activities, Adaptation & Aging. 2016/01/02 2016;40(1):1-19. doi:10.1080/01924788.2016.1127041
- [Background] Peters R, Ee N, Ward SA, Kenning G, Radford K, Goldwater M, Dodge HH, Lewis E, Xu Y, Kudrna G, Hamilton M, Peters J, Anstey KJ, Lautenschlager NT, Fitzgerald A, Rockwood K. Intergenerational Programmes bringing together community dwelling non-familial older adults and children: A Systematic Review. Arch Gerontol Geriatr. 2021 May-Jun;94:104356. doi: 10.1016/j.archger.2021.104356. Epub 2021 Jan 28. PMID 33567363
- [Background] Kim Y, Kim J, Lee JM, Seo DC, Jung HC. Intergenerational Taekwondo Program: A Narrative Review and Practical Intervention Proposal. Int J Environ Res Public Health. 2022 Apr 26;19(9):5247. doi: 10.3390/ijerph19095247. PMID 35564642
- [Background] Rizzo N. Fitness Industry Statistics 2021-2028 [Market Research]. 2021. https://runrepeat.com/fitness-industry
- [Background] Russell D, Peplau LA, Ferguson ML. Developing a measure of loneliness. J Pers Assess. 1978 Jun;42(3):290-4. doi: 10.1207/s15327752jpa4203_11. PMID 660402
- [Background] Koenig HG, Westlund RE, George LK, Hughes DC, Blazer DG, Hybels C. Abbreviating the Duke Social Support Index for use in chronically ill elderly individuals. Psychosomatics. 1993 Jan-Feb;34(1):61-9. doi: 10.1016/S0033-3182(93)71928-3. PMID 8426892
- [Background] Rikli RE, Jones CJ. Development and Validation of a Functional Fitness Test for Community-Residing Older Adults. Journal of Aging and Physical Activity. 01 Apr. 1999 1999;7(2):129-161. doi:10.1123/japa.7.2.129